CLINICAL TRIAL: NCT04026633
Title: Using Counter Attitudinal Advocacy to Change Drinking Behavior & Related Problems
Brief Title: Attitudes & College Experiences
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooklyn College of the City University of New York (Other)
Responsible Party: Principal Investigator, Angelo DiBello, Assistant Professor, Brooklyn College of the City University of New York
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AA025676 (NIH)
Record Dates: First submitted 2019-07-11; First posted 2019-07-19 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Abuse
Keywords: Alcohol Intervention; College Students
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Enhanced Intervention (Experimental): Participants assigned to this arm will complete a personal writing task about alcohol use.
  Interventions: Behavioral: CAA
- Placebo Comparator (Placebo Comparator): Participants assigned to this arm will complete a personal writing task about eating behaviors.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: CAA — Participants will write about the use of PBS and alcohol use.
  Arms: Experimental: Enhanced Intervention
Behavioral: Control — Participants will write about eating and exercise.
  Arms: Placebo Comparator

SUMMARY:
High volume drinking by young adults has proven resistant to long term change, so new approaches are needed. Given strong associations between alcohol-related attitudes and drinking behavior, the investigators adapt a theory-based attitude change strategy for use in alcohol prevention. This research tests the impact of a brief counter attitudinal advocacy activity on subsequent drinking and negative consequences.

DETAILED DESCRIPTION:
The persistence of risky drinking among young adults in college calls for continued efforts to prevent harms related to alcohol. Current prevention interventions have achieved some success, but rely on a single mechanism of change: correcting exaggerated drinking norms. The investigators propose to test a novel prevention strategy targeting another mechanism of change: creating attitude-behavior dissonance. To date, changing alcohol-related attitudes and the resulting attitude-behavior discrepancy has been underutilized as a behavior change strategy for alcohol abuse prevention. Informed by an extensive literature showing strong and consistent associations between alcohol attitudes and drinking behavior, the investigators adapted a brief counter-attitudinal advocacy (CAA) manipulation to the alcohol prevention context.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years of age
* Enrolled in the university's undergraduate four-year degree program
* Past month heavy episodic drinking (for men, >5 drinks in one day, for women >4 drinks in one day)
* At least two self-reported negative consequence from drinking in the past month

Exclusion Criteria:

• Status as a graduating senior

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Alcohol Consumption from Baseline to 1-Month | 1 month after baseline
  Average of reports from past 30 days on the number of standard drinks consumed by participant over the past 30 days.
Change in Alcohol-related consequences from Baseline to 1- and 3-Months | 1 month and 3 months after baseline
  The Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ) (Kahler et al., 2005) is a 24-item self-administered checklist of problems related to drinking; responses are dichotomous (yes/no) and refer to the past month which was collected at baseline and 5-months. The BYAACQ demonstrates strong psychometric properties and is free of gender bias (Kahler et al., 2005).

CONTACTS AND LOCATIONS:
Locations (1):
- Brooklyn College, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and the results of the study have been published, de-identified data will be made available to other qualified investigators upon request. The request will be evaluated by the investigators to ensure that it meets reasonable demands of scientific integrity.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Within one year of study completion
Access Criteria: To be determined